CLINICAL TRIAL: NCT04522648
Title: Prospective Surveillance for Breast Cancer-Related Lymphedema: A Randomized Trial
Brief Title: Prospective Surveillance for Breast Cancer-Related Lymphedema
Acronym: PROTECT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Rigshospitalet, Denmark (Other)
Collaborators: Aarhus University Hospital (Other); Odense University Hospital (Other); Zealand University Hospital (Other); Herlev Hospital (Other)
Responsible Party: Principal Investigator, Bolette Rafn, Postdoc, Rigshospitalet, Denmark
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: PROTECT
Record Dates: First submitted 2020-08-18; First posted 2020-08-21 (Actual); Last update posted 2023-08-18 (Actual); Status verified 2023-08

CONDITIONS: Breast Cancer
Keywords: lymphedema; Prospective surveillance
MeSH Terms: conditions — Breast Neoplasms; Lymphedema

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (INT) (Experimental): INT participants will be asked to perform self-measurements of arm circumference at five points along the arm at home every three months. Additional measurements can be performed if the participants experience signs of BCRL. Participants will report the self-measurements in cm and mm in an online questionnaire, or over the phone to a physiotherapist navigator, along with reporting sign and symptoms of BCRL.
  Interventions: Other: Prospective surveillance
- Control (CON) (No Intervention): The CON group will follow the usual post-operative care. CON participants will be prompted every 6 months by an online questionnaire to report if they have been diagnosed with BCRL and if so, month of initiation of treatment.

INTERVENTIONS:
Other: Prospective surveillance — A participant with an increase from pre-surgery in total arm volume of ≥6% by self-measurement, or symptoms of BCRL ≥2 NRS will receive an assessment by a lymphedema therapist. At this appointment, participants will receive a physical examination of the arm along with a BIS measurement. A participant is considered having subclinical BCRL if an increase in lymphedema index (L-DEX) ≥7 from pre-surgery measured by BIS is identified. A fitted compression garment and gauntlet is then provided, free of charge, for daily wear 10 hours/day for four weeks along with a recommendation to use the arm for daily activities and maintain regular physical activity. Following the four-week compression period, participants will be re-measured using BIS to evaluate response. Participants who do not respond to compression will receive CDT delivered by the lymphedema therapist.
  Arms: Intervention (INT)

SUMMARY:
This randomized trial will test the effect of a prospective surveillance program for early detection and subclinical management of breast cancer-related lymphedema on the prevalence of chronic lymphedema.

DETAILED DESCRIPTION:
Design and setting: This trial is a multi-center single-blind trial involving five hospitals in Denmark.

Procedure: All women booked for surgery for breast cancer at one of the study sites will be invited to participate. Women, who provide written informed consent, will have BIS measurements, and perform self-measurements of arm circumference. Further, participants will complete a sociodemographic questionnaire which will be used to ensure recruitment of a representable sample. This data will be collected at the hospital of surgery at pre-treatment. After surgery, women who had >6 lymph nodes removed and have planned radiation therapy will be randomized 1:1 into intervention or control.

ELIGIBILITY:
Inclusion Criteria:

* female;
* ≥18 years;
* surgery for breast cancer (unilateral and bilateral) including ALDN with >6 lymph nodes removed;
* can effectively communicate verbally in Danish;

Exclusion Criteria:

* surgery for breast cancer with SLNB or < 6 nodes removed;
* pre-existing lymphedema (primary or secondary);
* previous treatment for breast cancer;
* pace maker;
* conditions known to cause swelling (pregnancy, congestive heart failure, chronic/acute renal disease, cor pulmonale, nephrotic syndrome, nephrosis, liver failure or cirrhosis, pulmonary edema, and thrombophlebitis or deep vein thrombosis in the arms).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2021-01-04 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Prevalence of chronic lymphedema | At 24 months post-surgery
  A binary outcome (y/n) defined as BIS ≥10 from pre-surgery or outside normal range ±10

SECONDARY OUTCOMES:
Time-to-treatment | INT group: will be collected throughtout the study period. CON group: at 6, 12, 18 and 24 months post-surgery
  INT group: The time (weeks) from surgery to first elevated L-DEX score which triggers immediate treatment along with time (weeks) to resolution of BCRL from diagnosis. For CON: time from surgery to BCRL diagnosis, time from diagnosis to BCRL treatment, and time from initiation to termination of treatment
Health-related quality of life | pre-treatment, 6, 12, 18 and 24 months post-surgery
  This will be measured by the EQ-5D questionnaire
Arm function | pre-treatment, 6, 12, 18 and 24 months post-surgery
  This will be measured by the QuickDASH questionnaire

CONTACTS AND LOCATIONS:
Locations (3):
- Denmark (3):
  - Copenhagen University Hospital Rigshospitalet, Copenhagen
  - Herlev Hospital, Herlev
  - Odense University Hospital, Odense

IPD SHARING:
Plan to Share IPD: No